CLINICAL TRIAL: NCT01469013
Title: A Randomized, Double-Blind, Placebo-Controlled, Dose-Ranging, Parallel-Group, Phase 2 Study of Baricitinib (LY3009104) in Japanese Patients With Active Rheumatoid Arthritis on Background Methotrexate Therapy
Brief Title: Oral Baricitinib (LY3009104)Treatment in Japanese Participants With Active Rheumatoid Arthritis on Background Methotrexate Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 14116; I4V-JE-JADN (Other: Eli Lilly and Company)
Record Dates: First submitted 2011-11-08; First posted 2011-11-10 (Estimated); Results first posted 2018-11-01 (Actual); Last update posted 2019-09-20 (Actual); Status verified 2019-09

CONDITIONS: Arthritis, Rheumatoid
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Sugars; baricitinib; Methotrexate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Placebo (Placebo Comparator): 2 placebo capsules administered orally once daily for 12 weeks. Participants who complete this treatment arm will be randomized in a 1:1 ratio to either the 4-mg baricitinib or 8-mg baricitinib arms. Participants rerandomized to 8-mg baricitinib arm at Week12 will switch to 4-mg baricitinib once a day after the approval of protocol amendment (d) and will receive that switched dose until Week 64.
  The dosage form changed from capsule in treatment period (up to Week 12) to tablet in extension period (Week 13 to 64) per protocol amendment (b).
  Interventions: Drug: Placebo; Drug: Methotrexate
- 1-mg Baricitinib (LY3009104) (Experimental): 1 x 1-mg baricitinib capsule + 1 identical placebo capsule, both administered orally once daily for 12 weeks. Participants who complete this treatment arm will be randomized in a 1:1 ratio to either the 4-mg baricitinib or 8-mg baricitinib arms. Participants rerandomized to 8-mg baricitinib arm at Week 12 will switch to 4-mg baricitinib once a day after the approval of protocol amendment (d) and will receive that switched dose until Week 64.
  The dosage form changed from capsule in treatment period (up to Week 12) to tablet in extension period (Week 13 to 64) per protocol amendment (b).
  Interventions: Drug: Placebo; Drug: Baricitinib; Drug: Methotrexate
- 2-mg Baricitinib (LY3009104) (Experimental): 2 x 1-mg baricitinib capsules administered orally once daily for 12 weeks. Participants who complete this treatment arm will be randomized in a 1:1 ratio to either the 4-mg baricitinib or 8-mg baricitinib arms. Participants rerandomized to 8-mg baricitinib arm at Week 12 will switch to 4-mg baricitinib once a day after the approval of protocol amendment (d) and will receive that switched dose until Week 64.
  The dosage form changed from capsule in treatment period (up to Week 12) to tablet in extension period (Week 13 to 64) per protocol amendment (b).
  Interventions: Drug: Baricitinib; Drug: Methotrexate
- 4-mg Baricitinib (LY3009104) (Experimental): 1 x 4-mg baricitinib capsule + 1 identical placebo capsule, both administered orally once daily for 12 weeks. Participants who complete this 12-week period will remain on this treatment regimen in tablet form.
  Interventions: Drug: Placebo; Drug: Baricitinib; Drug: Methotrexate
- 8-mg Baricitinib (LY3009104) (Experimental): 2 x 4-mg baricitinib capsules administered orally once daily for 12 weeks. Participants who complete this 12-week period will remain on this treatment regimen in tablet form. Participants taking 8-mg baricitinib tablet form will switch to 4-mg baricitinib once a day after the approval of protocol amendment (d) and will receive that switched dose until Week 64.
  Interventions: Drug: Baricitinib; Drug: Methotrexate

INTERVENTIONS:
Drug: Placebo
  Other Names: Sugar pill
  Arms: 1-mg Baricitinib (LY3009104); 4-mg Baricitinib (LY3009104); Placebo
Drug: Baricitinib
  Other Names: JAK1/JAK2 inhibitor; JAK1 inhibitor; JAK2 inhibitor; NCB028050; LY3009104
  Arms: 8-mg Baricitinib (LY3009104)
Drug: Baricitinib
  Other Names: JAK1/JAK2 inhibitor; JAK1 inhibitor; JAK2 inhibitor; NCB028050; LY3009104
  Arms: 4-mg Baricitinib (LY3009104)
Drug: Baricitinib
  Other Names: JAK1/JAK2 inhibitor; JAK1 inhibitor; JAK2 inhibitor; NCB028050; LY3009104
  Arms: 1-mg Baricitinib (LY3009104); 2-mg Baricitinib (LY3009104); 4-mg Baricitinib (LY3009104); 8-mg Baricitinib (LY3009104)
Drug: Methotrexate — Administered orally as background therapy

SUMMARY:
This is a Phase 2b, outpatient, randomized, double-blinded (with a single-blind extension), placebo-controlled, dose-ranging, parallel-group study of baricitinib (LY3009104) in Japanese participants with active rheumatoid arthritis (RA) on background methotrexate (MTX) therapy. Baricitinib will be orally administered once a day with background methotrexate [6 to 16 milligrams (mg)/week] therapy for 12 weeks in the double-blind treatment period (1, 2, 4 or 8 mg/day, or placebo), and for 52 weeks in the single-blind extension period (4 or 8 mg/day).

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory males or females between the ages of 20 and 75 years, inclusive, at time of study entry
* Diagnosis of adult-onset RA (of at least 6 months duration but not longer than 15 years prior to screening) according to the 2010 American College of Rheumatology (ACR)/European League Against Rheumatism (EULAR) Responder Index classification criteria for RA
* Have active RA defined as at least 6 swollen and at least 6 tender joints based on the 66/68 joint count
* Regular use of MTX for at least 12 weeks, and treatment at a stable dose of 6 to 16 mg/week (2 or 3 times a week) for at least 8 weeks prior to the treatment period. The dose of MTX should remain stable throughout the study, but may be adjusted for safety reasons.
* For participants receiving corticosteroids, they must be on a dose not to exceed 10 mg of prednisone daily (or equivalent) and have been on the same dosing regimen for at least 6 weeks prior to the treatment period
* Have C-Reactive Protein (CRP) measurement > 0.5 milligrams/deciliter (mg/dL) or Erythrocyte Sedimentation Rate (ESR) > 28 millimeters/hour (mm/hr). The CRP and ESR may be repeated once during the screening period at the discretion of the investigator, and the repeat results may be accepted for study eligibility purposes

Exclusion Criteria:

* Use of nonsteroidal anti-inflammatories (NSAIDs) for less than 4 weeks prior to the treatment period. If on NSAIDs, must be on a stable dose of the drug for at least 4 weeks prior to the treatment period and must remain on a stable dose throughout the study
* Received prior treatment with an oral Janus Kinase (JAK) inhibitor regardless of when they received it
* Have a diagnosis of Felty's syndrome
* Evidence of human immunodeficiency virus (HIV) infection and/or positive human HIV antibodies
* Have hepatitis C virus (HCV; positive for anti-hepatitis C antibody with confirmed presence of HCV)
* Positive for hepatitis B surface antigen (HBsAg+), OR negative for hepatitis B surface antigen (HBsAg-), but positive for hepatitis B core antibody (HBcAb+) and/or positive for hepatitis B surface antibody (HBsAb+) with positive Hepatitis B virus (HBV)-deoxyribonucleic acid (DNA) [≥2.1 Log copy/mL by Polymerase Chain Reaction (PCR) method] detected in the serum
* Have a positive result of the QuantiFERON®-tuberculosis (TB) Gold test (QFT-G) or a purified protein derivative (PPD) test
* Have estimated Glomerular Filtration Rate (GFR) from serum creatinine using the Modification of Diet in Renal Disease (MDRD) method of <50 milliliter/minute (mL/min)

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2011-11; Primary Completion 2012-11 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (14):
- Japan (14):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chiba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fukuoka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hiroshima
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hokkaido
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hyōgo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ibaraki
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kagoshima
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kanagawa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nagasaki
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Okayama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Osaka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ōita
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tokyo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Toyama

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] Taylor PC, Takeuchi T, Burmester GR, Durez P, Smolen JS, Deberdt W, Issa M, Terres JR, Bello N, Winthrop KL. Safety of baricitinib for the treatment of rheumatoid arthritis over a median of 4.6 and up to 9.3 years of treatment: final results from long-term extension study and integrated database. Ann Rheum Dis. 2022 Mar;81(3):335-343. doi: 10.1136/annrheumdis-2021-221276. Epub 2021 Oct 27. PMID 34706874
- [Derived] Combe B, Balsa A, Sarzi-Puttini P, Tony HP, de la Torre I, Rogai V, Durand F, Witt S, Zhong J, Dougados M. Efficacy and safety data based on historical or pre-existing conditions at baseline for patients with active rheumatoid arthritis who were treated with baricitinib. Ann Rheum Dis. 2019 Aug;78(8):1135-1138. doi: 10.1136/annrheumdis-2018-214261. Epub 2019 Mar 6. No abstract available. PMID 30842122
- [Derived] Taylor PC, Kremer JM, Emery P, Zuckerman SH, Ruotolo G, Zhong J, Chen L, Witt S, Saifan C, Kurzawa M, Otvos JD, Connelly MA, Macias WL, Schlichting DE, Rooney TP, de Bono S, McInnes IB. Lipid profile and effect of statin treatment in pooled phase II and phase III baricitinib studies. Ann Rheum Dis. 2018 Jul;77(7):988-995. doi: 10.1136/annrheumdis-2017-212461. Epub 2018 Feb 20. PMID 29463520
- [Derived] Tanaka Y, Ishii T, Cai Z, Schlichting D, Rooney T, Macias W. Efficacy and safety of baricitinib in Japanese patients with active rheumatoid arthritis: A 52-week, randomized, single-blind, extension study. Mod Rheumatol. 2018 Jan;28(1):20-29. doi: 10.1080/14397595.2017.1307899. Epub 2017 Apr 25. PMID 28440680
- [Derived] Tanaka Y, Emoto K, Cai Z, Aoki T, Schlichting D, Rooney T, Macias W. Efficacy and Safety of Baricitinib in Japanese Patients with Active Rheumatoid Arthritis Receiving Background Methotrexate Therapy: A 12-week, Double-blind, Randomized Placebo-controlled Study. J Rheumatol. 2016 Mar;43(3):504-11. doi: 10.3899/jrheum.150613. Epub 2016 Feb 1. PMID 26834213

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants on background methotrexate therapy were assigned to a dose of 1, 2, 4, 8 mg baricitinib (LY3009104) or placebo capsule once daily in a double blind manner for 12 weeks followed by single blind treatment of 4 mg or 8 mg baricitinib (LY3009104) tablet once daily for 52 weeks extension period.
Groups:
- Part A: 1 mg Baricitinib (LY3009104): Participants on background methotrexate therapy administered 1 x 1-mg baricitinib (LY3009104) capsule + 1 identical placebo capsule, orally once daily for 12 weeks.
- Part A: 2 mg Baricitinib (LY3009104): Participants on background methotrexate therapy administered 2 x 1-mg baricitinib (LY3009104) capsules orally once daily for 12 weeks.
- Part A: 4 mg Baricitinib (LY3009104): Participants on background methotrexate therapy administered 1 x 4-mg baricitinib (LY3009104) capsule +1 identical placebo capsule, orally once daily for 12 weeks.
- Part A: 8 mg Baricitinib (LY3009104): Participants on background methotrexate therapy administered 2 x 4-mg baricitinib (LY3009104) capsules orally once daily for 12 weeks.
- Part A: Placebo: Participants on background methotrexate therapy administered 2 placebo capsules, orally once daily for 12 weeks.
- Part:1 mg Baricitinib(LY3009104) / 4 mg Baricitinib(LY3009104): Participants on background methotrexate therapy who were administered 1 x 1-mg LY3009104 capsule +1 identical placebo capsule, orally once daily for 12 weeks in Part A received 4 mg LY3009104 and 1 placebo tablet orally once daily for 52 weeks in Part B.
- Part B: 2 mg Baricitinib (LY3009104) / 4 mg Baricitinib (LY30: Participants on background methotrexate therapy who were administered 2 x 1-mg baricitinib (LY3009104) capsules orally once daily for 12 weeks in Part A received 4 mg baricitinib (LY3009104) and 1 placebo tablet orally once daily for 52 weeks in Part B.
- Part B: 4 mg Baricitinib (LY3009104) / 4 mg Baricitinib (LY30: Participants on background methotrexate therapy who were administered 1 x 4-mg baricitinib (LY3009104) capsule + 1 identical placebo capsule, orally once daily for 12 weeks in Part A received 4 mg baricitinib (LY3009104) and 1 placebo tablet orally once daily for 52 weeks in Part B.
- Part B: Placebo /4 mg Baricitinib (LY3009104): Participants on background methotrexate therapy who were administered 2 placebo capsules orally once daily for 12 weeks in Part A received 4 mg baricitinib (LY3009104) and 1 placebo tablet orally once daily for 52 weeks in Part B.
- Part B: 1 mg Baricitinib (LY3009104) / 8 mg Baricitinib (LY30: Participants on background methotrexate therapy who were administered 1 x 1-mg baricitinib (LY3009104) capsule + 1 identical placebo capsule orally once daily for 12 weeks in Part A received 2 x 4 mg baricitinib (LY3009104) tablets orally once daily for 52 weeks in Part B.
- Part B: 2 mg Baricitinib (LY3009104) / 8 mg Baricitinib (LY300: Participants on background methotrexate therapy who were administered 2 x 1-mg baricitinib (LY3009104) capsules orally once daily for 12 weeks in Part A received 2 x 4 mg baricitinib (LY3009104) tablets orally once daily for 52 weeks in Part B.
- Part B: 8 mg Baricitinib (LY3009104) / 8 mg Baricitinib (LY30: Participants on background methotrexate therapy who were administered 2 x 4-mg baricitinib (LY3009104) capsules orally once daily for 12 weeks in Part A received 2 x 4 mg baricitinib (LY3009104) tablets orally once daily for 52 weeks in Part B.
- Part B: Placebo / 8 mg Baricitinib (LY3009104): Participants on background methotrexate therapy who were administered 2 placebo capsules orally once daily for 12 weeks in Part A received 2 x 4 mg baricitinib (LY3009104) tablets orally once daily for 52 weeks in Part B.
Period: Part A (Treatment Period)
Arm/Group | Part A: 1 mg Baricitinib (LY3009104) | Part A: 2 mg Baricitinib (LY3009104) | Part A: 4 mg Baricitinib (LY3009104) | Part A: 8 mg Baricitinib (LY3009104) | Part A: Placebo | Part:1 mg Baricitinib(LY3009104) / 4 mg Baricitinib(LY3009104) | Part B: 2 mg Baricitinib (LY3009104) / 4 mg Baricitinib (LY30 | Part B: 4 mg Baricitinib (LY3009104) / 4 mg Baricitinib (LY30 | Part B: Placebo /4 mg Baricitinib (LY3009104) | Part B: 1 mg Baricitinib (LY3009104) / 8 mg Baricitinib (LY30 | Part B: 2 mg Baricitinib (LY3009104) / 8 mg Baricitinib (LY300 | Part B: 8 mg Baricitinib (LY3009104) / 8 mg Baricitinib (LY30 | Part B: Placebo / 8 mg Baricitinib (LY3009104)
Started | 24 | 24 | 24 | 24 | 49 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Received at Least 1 Dose of Study Drug | 24 | 24 | 24 | 24 | 49 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 23 | 24 | 23 | 24 | 48 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part B (Extension Period)
Arm/Group | Part A: 1 mg Baricitinib (LY3009104) | Part A: 2 mg Baricitinib (LY3009104) | Part A: 4 mg Baricitinib (LY3009104) | Part A: 8 mg Baricitinib (LY3009104) | Part A: Placebo | Part:1 mg Baricitinib(LY3009104) / 4 mg Baricitinib(LY3009104) | Part B: 2 mg Baricitinib (LY3009104) / 4 mg Baricitinib (LY30 | Part B: 4 mg Baricitinib (LY3009104) / 4 mg Baricitinib (LY30 | Part B: Placebo /4 mg Baricitinib (LY3009104) | Part B: 1 mg Baricitinib (LY3009104) / 8 mg Baricitinib (LY30 | Part B: 2 mg Baricitinib (LY3009104) / 8 mg Baricitinib (LY300 | Part B: 8 mg Baricitinib (LY3009104) / 8 mg Baricitinib (LY30 | Part B: Placebo / 8 mg Baricitinib (LY3009104)
Started | 0 | 0 | 0 | 0 | 0 | 12 | 12 | 23 | 24 | 11 | 12 | 24 | 24
Received at Least 1 Dose of Study Drug | 0 | 0 | 0 | 0 | 0 | 12 | 12 | 23 | 24 | 11 | 12 | 24 | 23 (1 participant discontinued prior to receiving study drug)
Completed | 0 | 0 | 0 | 0 | 0 | 10 | 7 | 18 | 20 | 8 | 10 | 18 | 18
Not Completed | 0 | 0 | 0 | 0 | 0 | 2 | 5 | 5 | 4 | 3 | 2 | 6 | 6
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 2 | 5 | 5 | 3 | 3 | 1 | 6 | 3
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 3

BASELINE CHARACTERISTICS:
Population: All randomized participants who received any amount of study treatment. All participants who completed Part A were re-randomized to 4 mg or 8 mg in Part B.
Groups:
- Part A: 1 mg Baricitinib (LY3009104): Participants on background methotrexate therapy were administered 1 mg baricitinib (LY3009104) orally once daily for 12 weeks in Part A and received 4 mg or 8 mg baricitinib (LY3009104) tablets orally once daily for 52 weeks in Part B.
- Part A: 2 mg Baricitinib (LY3009104): Participants on background methotrexate therapy were administered 2 mg baricitinib (LY3009104) orally once daily for 12 weeks in Part A and received 4 mg or 8 mg baricitinib (LY3009104) tablets orally once daily for 52 weeks in Part B.
- Part A: 4 mg Baricitinib (LY3009104): Participants on background methotrexate therapy were administered 4 mg baricitinib (LY3009104) orally once daily for 12 weeks in Part A and received 4 mg or 8 mg baricitinib (LY3009104) tablets orally once daily for 52 weeks in Part B.
- Part A: 8 mg Baricitinib (LY3009104): Participants on background methotrexate therapy were administered 8 mg baricitinib (LY3009104) orally once daily for 12 weeks in Part A and received 4 mg or 8 mg baricitinib (LY3009104) tablets orally once daily for 52 weeks in Part B.
- Part A: Placebo: Participants on background methotrexate therapy were administered placebo orally once daily for 12 weeks in Part A and received 4 mg or 8 mg baricitinib (LY3009104) tablets orally once daily for 52 weeks in Part B.
- Total: Total of all reporting groups
Arm/Group | Part A: 1 mg Baricitinib (LY3009104) | Part A: 2 mg Baricitinib (LY3009104) | Part A: 4 mg Baricitinib (LY3009104) | Part A: 8 mg Baricitinib (LY3009104) | Part A: Placebo | Total
Number analyzed (Participants) | 24 | 24 | 24 | 24 | 49 | 145
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.7 (12.8) | 56.1 (11.5) | 57.5 (10.4) | 53.6 (11.3) | 51.1 (12.0) | 53.6 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 21 | 19 | 17 | 39 | 118
  Male | 2 | 3 | 5 | 7 | 10 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 24 | 24 | 24 | 24 | 49 | 145
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 24 | 24 | 24 | 24 | 49 | 145
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 24 | 24 | 24 | 24 | 49 | 145

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants in the 4 mg and 8 mg Dose Groups Who Achieved an American College of Rheumatology 20 (ACR20) Responder Index Response Baseline Through Week 12 .
Description: ACR20 responders are participants with at least 20% improvement from baseline for tender joint count (TJC), swollen joint count (SJC), and at least 3 of the 5 remaining core set measures: Health Assessment Questionnaire-Disability Index (HAQ-DI) which measured participants perceived degree of difficulty performing daily activities, C-reactive Protein (CRP) and erythrocyte sedimentation rate (ESR), Patient's Assessment of Arthritis Pain-Visual Analog Scale (PAAP-VAS) , Patient's Global Assessment of Disease Activity-VAS (PtGADA-VAS), and Physician's Global Assessment of Disease Activity-VAS (PhGA-VAS). Missing values were imputed using Non-Responder Imputation (NRI), where non-responders were participants who discontinued the study prior to the completion of Part A. Percentage of participants achieving ACR20 response = (number of ACR20 responders) /(number of participants treated) * 100.
Time Frame: 12 weeks
Population: All participants who received at least 1 dose of 4 mg, 8 mg baricitinib (LY3009104) or placebo in Part A as per protocol for combined analysis .
Measure: Number; unit: percentage of participants
Groups:
- Part A: Combined 4 mg and 8 mg Baricitinib (LY3009104): Participants on background methotrexate therapy administered 1- 4 mg baricitinib (LY3009104) capsule +1 identical placebo capsule or 2 x 4-mg baricitinib (LY3009104) capsules, orally once daily for 12 weeks.
Arm/Group | Part A: Combined 4 mg and 8 mg Baricitinib (LY3009104) | Part A: Placebo
Number analyzed (Participants) | 48 | 49
percentage of participants | 77 | 31
Statistical Analysis 1: Comparison: Part A: Combined 4 mg and 8 mg Baricitinib (LY3009104) vs Part A: Placebo; Test type: Superiority or Other; p < 0.001, Regression, Logistic

2. Secondary Outcome: Percentage of Participants Who Achieved an ACR20 Response at 64 Weeks
Description: ACR20 responders are participants with at least 20% improvement from baseline for TJC, SJC, and at least 3 of the 5 remaining core set measures: HAQ-DI which measured participants perceived degree of difficulty performing daily activities, CRP and ESR, PAAP-VAS, PtGADA-VAS, or PhGA-VAS. Missing values were imputed using NRI, where non-responders were participants who discontinued the study prior to the completion of Part B. Percentage of participants achieving ACR20 response = (number of ACR20 responders) / (number of participants treated) * 100.
Time Frame: Baseline up to 64 weeks
Population: All participants who received any amount of study drug in Part B.
Measure: Number; unit: percentage of participants
Groups:
- Combined 4 mg Baricitinib (LY3009104) (Part B): Participants on background methotrexate therapy who were administered 1 mg, 2 mg, 4 mg baricitinib (LY3009104) capsule or placebo capsule, orally once daily for 12 weeks in Part A received 4 mg baricitinib (LY3009104) and 1 placebo tablet orally once daily for 52 weeks in Part B.
- Combined 8 mg Baricitinib (LY3009104) (Part B): Participants on background methotrexate therapy who were administered 1 mg, 2 mg, 8 mg baricitinib (LY3009104) capsule or placebo capsule, orally once daily for 12 weeks in Part A received 2 x 4 mg baricitinib (LY3009104) tablets orally once daily for 52 weeks in Part B.
Arm/Group | Combined 4 mg Baricitinib (LY3009104) (Part B) | Combined 8 mg Baricitinib (LY3009104) (Part B)
Number analyzed (Participants) | 71 | 70
percentage of participants | 66 | 73

3. Secondary Outcome: Percentage of Participants Who Achieved an ACR70 Response at 12 Weeks (Part A)
Description: ACR70 responders were participants with at least 70% improvement from baseline for TJC, SJC, and at least 3 of the 5 remaining core set measures: HAQ-DI, CRP, PAAP-VAS, PtGADA-VAS, or PhGA-VAS. Missing values were imputed using NRI, where non-responders were participants who discontinued the study prior to the completion of Part A. Percentage of participants achieving ACR70 response=(number of ACR70 responders / number of participants treated) * 100.
Time Frame: Baseline up to 12 weeks
Population: All participants who received any study drug in Part A.
Measure: Number; unit: percentage of participants
Groups:
- 1 mg Baricitinib (LY3009104): Participants on background methotrexate therapy administered 1 x 1-mg baricitinib (LY3009104) capsule + 1 identical placebo capsule, orally once daily for 12 weeks.
- 2 mg Baricitinib (LY3009104): Participants on background methotrexate therapy administered 2 x 1-mg baricitinib (LY3009104) capsules orally once daily for 12 weeks.
- 4 mg Baricitinib (LY3009104): Participants on background methotrexate therapy administered 1 x 4-mg baricitinib (LY3009104) capsule +1 identical placebo capsule, orally once daily for 12 weeks.
- 8 mg Baricitinib (LY3009104): Participants on background methotrexate therapy administered 2 x 4-mg baricitinib (LY3009104) capsules orally once daily for 12 weeks.
- Placebo: Participants on background methotrexate therapy administered 2 placebo capsules, orally once daily for 12 weeks.
Arm/Group | 1 mg Baricitinib (LY3009104) | 2 mg Baricitinib (LY3009104) | 4 mg Baricitinib (LY3009104) | 8 mg Baricitinib (LY3009104) | Placebo
Number analyzed (Participants) | 24 | 24 | 24 | 24 | 49
percentage of participants | 13 | 29 | 29 | 21 | 0
Statistical Analysis 1: Comparison: 1 mg Baricitinib (LY3009104) vs 2 mg Baricitinib (LY3009104) vs 4 mg Baricitinib (LY3009104) vs 8 mg Baricitinib (LY3009104) vs Placebo; Test type: Superiority or Other; p = 0.009, Cochran-Armitage trend test

4. Secondary Outcome: Percentage of Participants Who Achieved an ACR70 Response at 64 Weeks (Part B)
Description: ACR70 responders were participants with at least 70% improvement from baseline for TJC, SJC, and at least 3 of the 5 remaining core set measures: HAQ-DI, CRP, PAAP-VAS, PtGADA-VAS, or PhGA-VAS. Missing values were imputed using NRI, where non-responders were participants who discontinued the study prior to the completion of Part B. Percentage of participants achieving ACR70 response=(number of ACR70 responders) / (number of participants treated) * 100.
Time Frame: Baseline up to 64 weeks
Population: All participants who received any study drug in Part B.
Measure: Number; unit: percentage of participants
Groups:
- Combined 4 mg Baricitinib (LY3009104): Participants on background methotrexate therapy who were administered 1 mg, 2 mg, 4 mg baricitinib (LY3009104) capsule or identical placebo capsule, orally once daily for 12 weeks in Part A received 4 mg baricitinib (LY3009104) and 1 placebo tablet orally once daily for 52 weeks in Part B.
- Combined 8 mg Baricitinib (LY3009104): Participants on background methotrexate therapy who were administered 1 mg, 2 mg, 8 mg baricitinib (LY3009104) capsules orally once daily for 12 weeks in Part A received 2 x 4 mg baricitinib (LY3009104) tablets orally once daily for 52 weeks in Part B.
Arm/Group | Combined 4 mg Baricitinib (LY3009104) | Combined 8 mg Baricitinib (LY3009104)
Number analyzed (Participants) | 71 | 70
percentage of participants | 37 | 34

5. Secondary Outcome: Mean Change From Baseline to Week 12 in Disease Activity Score (DAS) Based on the 28 Diarthrodial Joint Count and CRP Level (DAS28-CRP)
Description: DAS modified included the DAS28 that consisted of a composite score of the following variables: tender joint count out of 28 (TJC28), swollen joint count out of 28 (SJC28), CRP [milligrams per liter (mg/L)], and PtGADA on a 0 to 100 millimeter (mm) VAS (0mm=no arthritis activity to 100 mm= extremely active arthritis). DAS28 calculated as: DAS28-CRP = 0.56(square root of TJC28)+0.28(square root of SJC28)+0.36[ln(CRP +1)]+0.014(VAS)+0.96. A decrease in DAS28-CRP indicated an improvement in participant's condition.
Time Frame: Baseline, 12 weeks
Population: All randomized participants who received any study drug in Part A and had DAS28-CRP evaluated at analysis time points. The last non-missing post-baseline value in Part A was used.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1 mg Baricitinib (LY3009104) | 2 mg Baricitinib (LY3009104) | 4 mg Baricitinib (LY3009104) | 8 mg Baricitinib (LY3009104) | Placebo
Number analyzed (Participants) | 24 | 24 | 24 | 24 | 49
units on a scale | -1.52 (0.970) | -2.02 (1.072) | -2.09 (1.105) | -1.96 (0.947) | -0.60 (1.204)

6. Secondary Outcome: Mean Change From Baseline to Week 64 in DAS Based on the 28 Diarthrodial Joint Count and CRP Level (DAS28-CRP)
Description: DAS modified included the 28 diarthroidal joint count (DAS28) that consisted of a composite score of the following variables: TJC28, SJC28, CRP (mg/L), and PtGADA on a 0 to 100 mm VAS (0mm=no arthritis activity to 100 mm= extremely active arthritis). DAS28 calculated as: DAS28-CRP = 0.56(square root of TJC28)+0.28(square root of SJC28)+0.36[ln(CRP +1)]+0.014(VAS)+0.96. A decrease in DAS28-CRP indicated an improvement in participant's condition.
Time Frame: Baseline, 64 weeks
Population: All randomized participants who received any study drug in Part B and had DAS28-CRP evaluated at analysis time points. The last non-missing post-baseline value in Part B was used.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Combined 4 mg Baricitinib (LY3009104) | Combined 8 mg Baricitinib (LY3009104)
Number analyzed (Participants) | 71 | 70
units on a scale | -2.44 (1.152) | -2.48 (1.109)

7. Secondary Outcome: Percentage of Participants Who Achieved an European League Against Rheumatism Rating of 28-Joint Arthritic Condition (EULAR28) Response at 12 Weeks (Part A)
Description: EULAR Responder Index based on 28 joint counts categorizes clinical response based on improvement from baseline in DAS28-CRP. DAS28-CRP scores range from 1.0-9.4, where lower scores indicated less disease activity. High disease activity: DAS28-CRP >5.1, low disease activity: DAS28-CRP ≤3.2, and remission: DAS28-CRP <2.6. Participants are categorized as EULAR responders or non-responders based on improvement of DAS28-CRP scores from baseline. EULAR DAS28-CRP responder index defines a good (absolute: ≤3.2 and >1.2 improvement from baseline), moderate (absolute: >3.2 and ≤5.1 and >0.6 and ≤1.2 improvement from baseline), or no response (absolute: >5.1 and ≤0.6 improvement from baseline). Percentage of participants calculated as = (number of good +moderate responders) / (number of participants treated) * 100.
Time Frame: Baseline up to 12 weeks
Population: All participants who received any amount of study drug in Part A.
Measure: Number; unit: percentage of participants
Arm/Group | 1 mg Baricitinib (LY3009104) | 2 mg Baricitinib (LY3009104) | 4 mg Baricitinib (LY3009104) | 8 mg Baricitinib (LY3009104) | Placebo
Number analyzed (Participants) | 24 | 24 | 24 | 24 | 49
percentage of participants | 83 | 88 | 92 | 92 | 47

8. Secondary Outcome: Percentage of Participants Who Achieved an EULAR28 Response at 64 Weeks (Part B)
Description: EULAR Responder Index based on 28 joint counts categorizes clinical response based on improvement from baseline in DAS28-CRP. DAS28-CRP scores range from 1.0-9.4, where lower scores indicated less disease activity. High disease activity: DAS28-CRP >5.1, low disease activity: DAS28-CRP <3.2, and remission: DAS28-CRP <2.6. Participants are categorized as EULAR responders or non-responders based on improvement of DAS28-CRP scores from baseline. EULAR DAS28-CRP Responder Index defines a good (absolute: ≤3.2 and >1.2 improvement from baseline), moderate (absolute: >3.2 and ≤5.1 and >0.6 and ≤1.2 improvement from baseline), or no response (absolute: >5.1 and ≤0.6 improvement from baseline). Percentage of participants calculated as = (number of good +moderate responders) / (number of participants treated) * 100.
Time Frame: Baseline up to 64 weeks
Population: All participants who received any amount of study drug in Part B.
Measure: Number; unit: percentage of participants
Arm/Group | Combined 4 mg Baricitinib (LY3009104) | Combined 8 mg Baricitinib (LY3009104)
Number analyzed (Participants) | 71 | 70
percentage of participants | 94 | 94

9. Secondary Outcome: Mean Change in Simplified Disease Activity Index (SDAI) Responses up to 12 Weeks (Part A)
Description: The SDAI is the numerical sum of 5 outcome parameters: TJC28, SJC28, patient and physician global assessment of disease activity and CRP. The equation used to calculate the SDAI:SDAI=SJC28+TJC28+PtGADA-VAS+PhGA-VAS+CRP where PtGADA-VAS=PtGADA-VAS / 10 and PhGA-VAS=PhGA-VAS / 10, with lower values indicating fewer symptoms.
Time Frame: Baseline up to 12 weeks
Population: All participants who received any amount of study drug in Part A and had SDAI data at analysis time points. The last non-missing post-baseline value in Part A was used.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1 mg Baricitinib (LY3009104) | 2 mg Baricitinib (LY3009104) | 4 mg Baricitinib (LY3009104) | 8 mg Baricitinib (LY3009104) | Placebo
Number analyzed (Participants) | 24 | 24 | 24 | 24 | 49
units on a scale | -13.11 (8.918) | -16.85 (9.517) | -18.17 (9.202) | -18.02 (8.293) | -4.54 (13.113)

10. Secondary Outcome: Mean Change in SDAI Responses up to 64 Weeks (Part B)
Description: The SDAI is the numerical sum of 5 outcome parameters: TJC28, SJC28, PtGADA, PhGA, and CRP. The equation used to calculate the SDAI:
  SDAI=SJC28+TJC28+PtGADA-VAS+PhGA-VAS+CRP where PtGADA-VAS=PtGADA -VAS/ 10 and PhGA-VAS=PhGA-VAS/ 10, with lower values indicating fewer symptoms.
Time Frame: Baseline, 64 weeks
Population: All participants who received any amount of study drug in Part B and had data for SDAI at analysis time points. The last non-missing post-baseline value in Part B was used.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Combined 4 mg Baricitinib (LY3009104) | Combined 8 mg Baricitinib (LY3009104)
Number analyzed (Participants) | 71 | 70
units on a scale | -20.42 (9.671) | -21.33 (10.318)

11. Secondary Outcome: Mean Change in Health Assessment Questionnaire - Disability Index (HAQ-DI) Responses up to 12 Weeks (Part A)
Description: HAQ-DI was a participant-reported questionnaire that consisted of 24 questions referring to 8 domains: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and daily activities. Participants assessed their ability to do each task over the week using response categories: without any difficulty (0), with some difficulty (1), with much difficulty (2), and unable to do (3). The highest score for any question in a category was the score of that category unless special aids or devices or help from another person was required. Answers for at least 6 of the 8 domains were required. Otherwise, HAQ-DI score was considered missing. The HAQ-DI score was the sum of the category scores divided by the number of categories scored, with a possible scores range from 0 to 3, 0 being without any difficulty and 3 being unable to do.
Time Frame: Baseline, 12 weeks
Population: All participants who received any amount of study drug in Part A and had HAQ-DI evaluated at analysis time points. The last non-missing post-baseline value in Part A was used.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1 mg Baricitinib (LY3009104) | 2 mg Baricitinib (LY3009104) | 4 mg Baricitinib (LY3009104) | 8 mg Baricitinib (LY3009104) | Placebo
Number analyzed (Participants) | 24 | 24 | 24 | 24 | 49
units on a scale | -0.302 (0.3336) | -0.396 (0.4759) | -0.469 (0.3463) | -0.422 (0.3646) | -0.077 (0.3552)

12. Secondary Outcome: Mean Change in HAQ-DI Responses up to 64 Weeks (Part B)
Description: HAQ-DI was a participant-reported questionnaire that consisted of 24 questions referring to 8 domains: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and daily activities. Participants assessed their ability to do each task over the week using response categories: without any difficulty (0); with some difficulty (1); with much difficulty (2); and unable to do (3). The highest score for any question in a category was the score of that category unless special aids or devices or help from another person was required. Answers for at least 6 of the 8 domains were required. Otherwise, HAQ-DI score was considered missing. The HAQ-DI score was the sum of the category scores divided by the number of categories scored, with a possible scores range from 0 to 3, 0 being without any difficulty and 3 being unable to do.
Time Frame: Baseline, 64 weeks
Population: All participants who received any amount of study drug in Part B and had HAQ-DI evaluated at analysis time points. The last non-missing post-baseline value in Part B was used.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Combined 4 mg Baricitinib (LY3009104) | Combined 8 mg Baricitinib (LY3009104)
Number analyzed (Participants) | 71 | 70
units on a scale | -0.498 (0.4779) | -0.568 (0.6203)

13. Secondary Outcome: Mean Value of ACR-N Response (Part A)
Description: The ACR-N Response Index is a continuous measure of clinical, laboratory, and functional measures in RA to characterize the percentage of improvement from baseline in RA disease activity. This index is defined as the lowest of either: a) percent change in TJC, b) percent change in SJC, or c) median percent change of the remaining 5 ACR core criteria (HAQ-DI, CRP, PAAP-VAS, PtGADA-VAS, or PhGA-VAS). A participant with an ACR-N of "X" has improvement of at least "X%" in tender and swollen joints and a median improvement of at least "X%" in the 5 remaining ACR core criteria. Since ACR-N is a continuous measure, the mean values are reported instead of the originally registered percentage of participants.
Time Frame: Baseline up to 12 weeks
Population: All participants who received any study drug in Part A and had baseline and at least one post baseline ACR-N response measure. LOCF was used to impute missing post-baseline values.
Measure: Mean (Standard Deviation); unit: percentage of responders
Groups:
- 8 mg Baricitinib (LY3009104): Participants on background methotrexate therapy administered 2 x 4-mg baricitinib (LY3009104) 4 capsules orally once daily for 12 weeks.
Arm/Group | 1 mg Baricitinib (LY3009104) | 2 mg Baricitinib (LY3009104) | 4 mg Baricitinib (LY3009104) | 8 mg Baricitinib (LY3009104) | Placebo
Number analyzed (Participants) | 23 | 24 | 23 | 24 | 48
percentage of responders | 28.76 (38.65) | 42.48 (39.52) | 45.17 (33.75) | 25.58 (130.02) | -9.98 (58.10)

14. Secondary Outcome: Mean Value of ACR-N Response (Part B)
Description: as for outcome 13
Time Frame: Baseline up to 64 weeks
Population: All participants who received any study drug in Part B and had baseline and at least one post baseline ACR-N response measure. LOCF was used to impute missing post-baseline values.
Measure: Mean (Standard Deviation); unit: percentage of responders
Arm/Group | Combined 4 mg Baricitinib (LY3009104) | Combined 8 mg Baricitinib (LY3009104)
Number analyzed (Participants) | 55 | 54
percentage of responders | 61.14 (30.70) | 61.07 (33.22)

15. Secondary Outcome: Percentage of Participants Who Achieved a DAS28 Remission at 12 Weeks (Part A)
Description: DAS modified included the DAS28 that consisted of a composite score of the following variables: TJC28, SJC28, CRP (mg/L), and PtGADA on a 0 to 100 mm VAS: 0 mm (no arthritis activity) to 100 mm (extremely active arthritis). DAS28 calculated as: DAS28-CRP = 0.56(square root of TJC28)+0.28(square root of SJC28)+0.36[ln(CRP +1)]+0.014(VAS)+0.96. For remission, DAS28 is <2.6. Percentage of participants = (number of participants with DAS28 remission) / (number of participants treated) * 100.
Time Frame: Baseline up to 12 weeks
Population: All participants who received any amount of study treatment in Part A.
Measure: Number; unit: percentage of participants
Arm/Group | 1 mg Baricitinib (LY3009104) | 2 mg Baricitinib (LY3009104) | 4 mg Baricitinib (LY3009104) | 8 mg Baricitinib (LY3009104) | Placebo
Number analyzed (Participants) | 24 | 24 | 24 | 24 | 49
percentage of participants | 33 | 33 | 42 | 50 | 22

16. Secondary Outcome: Percentage of Participants Who Achieved a DAS28 Remission at 64 Weeks (Part B)
Description: DAS modified included the DAS28 that consisted of a composite score of the following variables: TJC28, SJC28, CRP (mg/L), and PtGADA-VAS on a 0 to 100 mm VAS: 0 mm (no arthritis activity) to 100 mm (extremely active arthritis). DAS28 calculated as: DAS28-CRP = 0.56(sqrt of TJC28)+0.28(sqrt of SJC28)+0.36[ln(CRP +1)]+0.014(VAS)+0.96. For remission, DAS28 is <2.6. Percentage of participants = (number of participants with DAS 28 remission) / (number of participants treated) * 100.
Time Frame: Baseline up to 64 weeks
Population: All participants who received any amount of study drug in Part B.
Measure: Number; unit: percentage of participants
Arm/Group | Combined 4 mg Baricitinib (LY3009104) | Combined 8 mg Baricitinib (LY3009104)
Number analyzed (Participants) | 71 | 70
percentage of participants | 66 | 66

17. Secondary Outcome: Percentage of Participants Who Achieved an SDAI Remission at 12 Weeks (Part A)
Description: The SDAI is the numerical sum of 5 outcome parameters: TJC28, SJC28, PtGADA, PhGA and CRP. The equation used to calculate the SDAI:
  SDAI=SJC28+TJC28+PtGADA-VAS+PhGA-VAS+CRP where PtGADA-VAS=PtGADA -VAS/ 10 and PhGA-VAS=PhGA-VAS / 10. Definition of remission is SDAI ≤ 3.3. Percentage of participants = (number of responders) / (number of participants treated) * 100
Time Frame: Baseline up to 12 weeks
Population: All participants who received any amount of study drug in Part A.
Measure: Number; unit: percentage of participants
Arm/Group | 1 mg Baricitinib (LY3009104) | 2 mg Baricitinib (LY3009104) | 4 mg Baricitinib (LY3009104) | 8 mg Baricitinib (LY3009104) | Placebo
Number analyzed (Participants) | 24 | 24 | 24 | 24 | 49
percentage of participants | 4 | 29 | 17 | 17 | 8

18. Secondary Outcome: Percentage of Participants Who Achieved an SDAI Remission at 64 Weeks (Part B)
Description: The SDAI is the numerical sum of 5 outcome parameters: TJC28, SJC28, PtGADA, PhGA, and CRP. The equation used to calculate the SDAI:
  SDAI=SJC28+TJC28+PtGADA-VAS+PhGA-VAS+CRP where PtGADA-VAS=PtGADA-VAS / 10 and PhGA-VAS=PhGA-VAS / 10. Definition of remission is SDAI ≤ 3.3. Percentage of participants = (number of responders) / (number of participants treated) * 100
Time Frame: Baseline up to 64 weeks
Population: All participants who received any amount of study drug in Part B.
Measure: Number; unit: percentage of participants
Arm/Group | Combined 4 mg Baricitinib (LY3009104) | Combined 8 mg Baricitinib (LY3009104)
Number analyzed (Participants) | 71 | 70
percentage of participants | 39 | 39

19. Secondary Outcome: Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve at a Dosing Interval at Steady State (AUCtau,ss) of LY3009104
Description: Steady state is achieved when the rate of drug input is equal to the rate of drug elimination. The AUC(tau,ss) at 1 dosing interval is the average concentration of the drug at steady state multiplied by the time of the dosing interval.
Time Frame: Weeks (Wks) 0, 8, 12, or 20: Predose, 15 to 30 minutes and 1 to 3 hours postdose; Wks 2 or 4 and 15 or 16: Predose; Wks 28, 40, 52, or 64: random single sample.
Population: All participants who received any study drug and had evaluable data for AUC(tau,ss).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomoles*hour (nM*h)
Arm/Group | 1 mg Baricitinib (LY3009104) | 2 mg Baricitinib (LY3009104) | 4 mg Baricitinib (LY3009104) | 8 mg Baricitinib (LY3009104)
Number analyzed (Participants) | 24 | 24 | 48 | 47
nanomoles*hour (nM*h) | 237 (28.8) | 525 (21) | 1020 (32.5) | 1900 (24.1)

20. Secondary Outcome: PK: Maximum Concentration at Steady State of Dosing (Cmax,ss) of LY3009104
Time Frame: Wks 0, 8, 12, or 20: Predose, 15 to 30 minutes and 1 to 3 hours postdose; Wks 2 or 4 and 15 or 16: Predose; Wks 28, 40, 52, or 64: random single sample.
Population: All participants who received any study drug and had evaluable Cmax data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM
Arm/Group | 1 mg Baricitinib (LY3009104) | 2 mg Baricitinib (LY3009104) | 4 mg Baricitinib (LY3009104) | 8 mg Baricitinib (LY3009104)
Number analyzed (Participants) | 24 | 24 | 48 | 47
nM | 35.7 (20.9) | 73.5 (22.5) | 147 (20.6) | 278 (21.7)

ADVERSE EVENTS:
Groups:
- Placebo / 4 mg Baricitinib (LY3009104): Participants on background methotrexate therapy who were administered placebo capsule, orally once daily for 12 weeks in Part A received 4 mg baricitinib (LY3009104) and 1 placebo tablet orally once daily for 52 weeks in Part B.
- 1 mg Baricitinib (LY3009104) / 4mg Baricitinib (LY3009104): Participants on background methotrexate therapy who were administered 1 mg baricitinib (LY3009104) capsule, orally once daily for 12 weeks in Part A received 4 mg baricitinib (LY3009104) and 1 placebo tablet orally once daily for 52 weeks in Part B.
- 2 mg Baricitinib (LY3009104) / 4 mg Baricitinib (LY3009104): Participants on background methotrexate therapy who were administered 2 mg baricitinib (LY3009104) capsule, orally once daily for 12 weeks in Part A received 4 mg baricitinib (LY3009104) and 1 placebo tablet orally once daily for 52 weeks in Part B.
- 4 mg Baricitinib (LY3009104) / 4 mg Baricitinib (LY3009104): Participants on background methotrexate therapy who were administered 4 mg baricitinib (LY3009104) capsule, orally once daily for 12 weeks in Part A received 4 mg baricitinib (LY3009104) and 1 placebo tablet orally once daily for 52 weeks in Part B.
- Placebo /8 mg Baricitinib (LY3009104): Participants on background methotrexate therapy who were administered placebo capsule, orally once daily for 12 weeks in Part A received 2 x 4 mg baricitinib (LY3009104) tablets orally once daily for 52 weeks in Part B.
- 1 mg Baricitinib (LY3009104) / 8 mg Baricitinib (LY3009104): Participants on background methotrexate therapy who were administered 1 mg baricitinib (LY3009104) capsule, orally once daily for 12 weeks in Part A received 2 x 4 mg baricitinib (LY3009104) tablets orally once daily for 52 weeks in Part B.
- 2 mg Baricitinib (LY3009104) / 8 mg Baricitinib (LY3009104): Participants on background methotrexate therapy who were administered 2 mg baricitinib (LY3009104) capsule, orally once daily for 12 weeks in Part A received 2 x 4 mg baricitinib (LY3009104) tablets orally once daily for 52 weeks in Part B.
- 8 mg Baricitinib (LY3009104) / 8 mg Baricitinib (LY3009104): Participants on background methotrexate therapy who were administered 8 mg baricitinib (LY3009104) capsule, orally once daily for 12 weeks in Part A received 2 x 4 mg baricitinib (LY3009104) tablets orally once daily for 52 weeks in Part B.
Arm/Group | Placebo | 1 mg Baricitinib (LY3009104) | 2 mg Baricitinib (LY3009104) | 4 mg Baricitinib (LY3009104) | 8 mg Baricitinib (LY3009104) | Placebo / 4 mg Baricitinib (LY3009104) | 1 mg Baricitinib (LY3009104) / 4mg Baricitinib (LY3009104) | 2 mg Baricitinib (LY3009104) / 4 mg Baricitinib (LY3009104) | 4 mg Baricitinib (LY3009104) / 4 mg Baricitinib (LY3009104) | Placebo /8 mg Baricitinib (LY3009104) | 1 mg Baricitinib (LY3009104) / 8 mg Baricitinib (LY3009104) | 2 mg Baricitinib (LY3009104) / 8 mg Baricitinib (LY3009104) | 8 mg Baricitinib (LY3009104) / 8 mg Baricitinib (LY3009104)
Serious Adverse Events (participants affected / at risk) | 1/49 | 0/24 | 1/24 | 0/24 | 1/24 | 1/24 | 1/12 | 3/12 | 3/23 | 2/23 | 2/11 | 2/12 | 6/24
Other Adverse Events (participants affected / at risk) | 26/49 | 11/24 | 12/24 | 13/24 | 17/24 | 21/24 | 11/12 | 11/12 | 22/23 | 23/23 | 11/11 | 12/12 | 23/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=49) | 1 mg Baricitinib (LY3009104) (N=24) | 2 mg Baricitinib (LY3009104) (N=24) | 4 mg Baricitinib (LY3009104) (N=24) | 8 mg Baricitinib (LY3009104) (N=24) | Placebo / 4 mg Baricitinib (LY3009104) (N=24) | 1 mg Baricitinib (LY3009104) / 4mg Baricitinib (LY3009104) (N=12) | 2 mg Baricitinib (LY3009104) / 4 mg Baricitinib (LY3009104) (N=12) | 4 mg Baricitinib (LY3009104) / 4 mg Baricitinib (LY3009104) (N=23) | Placebo /8 mg Baricitinib (LY3009104) (N=23) | 1 mg Baricitinib (LY3009104) / 8 mg Baricitinib (LY3009104) (N=11) | 2 mg Baricitinib (LY3009104) / 8 mg Baricitinib (LY3009104) (N=12) | 8 mg Baricitinib (LY3009104) / 8 mg Baricitinib (LY3009104) (N=24)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Meniere's disease (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Forearm fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ulna fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Viith nerve paralysis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Placebo (N=49) | 1 mg Baricitinib (LY3009104) (N=24) | 2 mg Baricitinib (LY3009104) (N=24) | 4 mg Baricitinib (LY3009104) (N=24) | 8 mg Baricitinib (LY3009104) (N=24) | Placebo / 4 mg Baricitinib (LY3009104) (N=24) | 1 mg Baricitinib (LY3009104) / 4mg Baricitinib (LY3009104) (N=12) | 2 mg Baricitinib (LY3009104) / 4 mg Baricitinib (LY3009104) (N=12) | 4 mg Baricitinib (LY3009104) / 4 mg Baricitinib (LY3009104) (N=23) | Placebo /8 mg Baricitinib (LY3009104) (N=23) | 1 mg Baricitinib (LY3009104) / 8 mg Baricitinib (LY3009104) (N=11) | 2 mg Baricitinib (LY3009104) / 8 mg Baricitinib (LY3009104) (N=12) | 8 mg Baricitinib (LY3009104) / 8 mg Baricitinib (LY3009104) (N=24)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 3 (4) | 3 (4) | 1 (1) | 1 (1) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Birth mark (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Deafness neurosensory (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thyroid mass (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thyroiditis (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thyroiditis chronic (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry eye (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aphthous stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cheilitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 1 (1)
Dental caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric polyps (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1)
Gastritis atrophic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastritis erosive (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hyperchlorhydria (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Pancreatitis chronic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Periodontal disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (4)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mass (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gallbladder polyp (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic cyst (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 3 (3) | 1 (2) | 2 (2) | 1 (1) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hepatic steatosis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Liver injury (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Allergy to arthropod sting (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bacteriuria (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eczema impetiginous (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Empyema (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Enteritis infectious (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Enterocolitis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Folliculitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fungal paronychia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fungal skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Furuncle (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (2)
Gastroenteritis norovirus (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Genital herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gingivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Helicobacter infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Herpes simplex (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Influenza (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Molluscum contagiosum (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 6 (7) | 2 (2) | 2 (2) | 2 (2) | 2 (2) | 4 (4) | 5 (6) | 6 (6) | 7 (8) | 9 (15) | 1 (1) | 1 (2) | 5 (9)
Oesophageal candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Paronychia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Periodontitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pertussis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 2 (6) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulpitis dental (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Skin candida (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinea pedis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tinea versicolour (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral rash (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vulval abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthropod sting (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chillblains (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lip injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sternal fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Blood cholesterol increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 4 (4) | 1 (1) | 0 (0) | 3 (3) | 4 (5) | 2 (2) | 2 (3) | 2 (2)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheterisation cardiac (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cell marker increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Colonoscopy (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Electrocardiogram st-t segment abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Endoscopy (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eosinophil count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Glomerular filtration rate decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic enzyme abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lipids abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Liver function test abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Low density lipoprotein increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophagogastroduodenoscopy (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transaminases increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Dyslipidaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 2 (2) | 1 (1) | 0 (0) | 3 (3)
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 2 (2) | 1 (1) | 3 (3)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyogenic granuloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cubital tunnel syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness postural (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Hyposmia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intercostal neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Visual field defect (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anxiety disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysphoria (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Head banging (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertonic bladder (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leukocyturia (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal cyst (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal impairment (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Dysmenorrhoea (Reproductive system and breast disorders) | 0/39 (0) | 0/22 (0) | 0/21 (0) | 0/19 (0) | 0/17 (0) | 0/21 (0) | 1/10 (1) | 0/9 (0) | 0/18 (0) | 0/17 (0) | 0 (0) | 0 (0) | 0/17 (0)
Menstrual disorder (Reproductive system and breast disorders) | 1/39 (1) | 0/22 (0) | 0/21 (0) | 0/19 (0) | 0/17 (0) | 0/21 (0) | 0/10 (0) | 0/9 (0) | 0/18 (0) | 0/17 (0) | 0 (0) | 0 (0) | 0/17 (0)
Ovarian cyst (Reproductive system and breast disorders) | 0/39 (0) | 0/22 (0) | 0/21 (0) | 0/19 (0) | 0/17 (0) | 0/21 (0) | 0/10 (0) | 1/9 (1) | 0/18 (0) | 1/17 (1) | 0 (0) | 0 (0) | 0/17 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 1 (2) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (3) | 1 (1) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acne cystic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (3) | 0 (0) | 0 (0) | 1 (1)
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Miliaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Xanthoma (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholecystectomy (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coronary angioplasty (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Drug delivery device implantation (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
External fixation of fracture (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal endoscopic therapy (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Internal fixation of fracture (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intraocular lens implant (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Medical device removal (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Open reduction of fracture (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Removal of foreign body (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tooth extraction (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound treatment (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Phlebitis (Vascular disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Varicose vein (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days